CLINICAL TRIAL: NCT07392021
Title: The Effects of a Recovery-Promoting Program on Self-Efficacy, Quality of Recovery, and Clinical Outcomes in Patients Undergoing Coronary Artery Bypass Graft Surgery
Brief Title: Effects of a Recovery-Promoting Program in Patients Undergoing CABG Surgery
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mahidol University (Other)
Collaborators: The Princess Mantarop Kamalas Foundation, The Nurses' Association of Thailand (Unknown); Ramathibodi School of Nursing, Mahidol University (Unknown)
Responsible Party: Principal Investigator, Thanyaphat Chaisunthararat, Registered Nurse and Graduate Student (Master of Nursing Science), Mahidol University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: COA.No.MURA2025/476, 148/2568; TCTR20250915012 (Registry Identifier: Thai Clinical Trials Registry)
Record Dates: First submitted 2026-01-21; First posted 2026-02-06 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Coronary Artery Disease (CAD); Coronary Artery Bypass Graft (CABG); Postoperative Recovery
Keywords: Coronary Artery Bypass Graft; Quality of Recovery; Enhanced Recovery After Cardiac Surgery; Self-Efficacy; Cardiac Rehabilitation; Pulmonary Function; Functional Capacity
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Intervention Model Description: This study uses a parallel-group design comparing two groups of patients undergoing coronary artery bypass graft surgery. Participants in the control group receive standard postoperative care, while participants in the experimental group receive a recovery-promoting program in addition to standard care. Outcomes are assessed and compared between groups at predefined time points.
Masking Description: This is an open-label study. No masking is applied to participants, care providers, investigators, or outcome assessors.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Recovery Promotion Program for CABG patients (Experimental): Participants in this arm receive an integrated recovery promotion program combining Cardiac Rehabilitation (CR) and Enhanced Recovery After Cardiac Surgery (ERAS) in addition to standard postoperative care. The program includes structured education, early mobilization, breathing exercises, symptom monitoring, and self-management support delivered by nurses through in-hospital sessions and a LINE Official Account after discharge. The intervention aims to enhance self-efficacy, promote functional recovery, and reduce postoperative complications following coronary artery bypass grafting (CABG).
  Interventions: Behavioral: Recovery Promotion Program for CABG patients
- Standard CABG Care (Active Comparator): Participants in this arm receive standard postoperative care according to hospital protocols for patients undergoing coronary artery bypass grafting (CABG). This includes routine medical and nursing care, usual postoperative monitoring, discharge education, and follow-up appointments without the structured integrated Cardiac Rehabilitation and ERAS program or LINE-based support.
  Interventions: Other: Standard Postoperative CABG Care

INTERVENTIONS:
Behavioral: Recovery Promotion Program for CABG patients — An integrated recovery promotion program combining Cardiac Rehabilitation (CR) and Enhanced Recovery After Cardiac Surgery (ERAS) principles. The intervention is delivered by trained nurses and physiotherapists and consists of three phases: (1) preoperative phase including patient education, breathing exercises, and psychological preparation; (2) postoperative in-hospital phase including early mobilization, pulmonary rehabilitation, symptom monitoring, and individualized guidance; and (3) post-discharge phase including weekly follow-up, self-management support, and remote monitoring via LINE Official Account for six weeks. The program is designed to enhance self-efficacy, promote functional recovery, and reduce postoperative complications following CABG.
  Arms: Recovery Promotion Program for CABG patients
Other: Standard Postoperative CABG Care — Standard postoperative care for patients undergoing coronary artery bypass grafting (CABG) according to Rajavithi Hospital protocols. Care includes routine medical and nursing care, postoperative monitoring, physiotherapy, medication management, discharge education, and scheduled follow-up without the structured integrated CR-ERAS program or tele-nursing support.
  Arms: Standard CABG Care

SUMMARY:
Patients undergoing coronary artery bypass graft (CABG) surgery often experience physical limitations, psychological stress, and challenges during recovery after hospital discharge. Inadequate preparation and limited follow-up support may affect patients' confidence in self-care and overall recovery.

The purpose of this study is to evaluate the effects of a recovery-promoting program on self-efficacy, quality of recovery, and clinical outcomes in patients undergoing CABG surgery.

Participants will receive standard postoperative care. In addition, participants in the intervention group will receive a recovery-promoting program provided by nurses, which includes structured education, guidance on postoperative activity and symptom management, and follow-up support after discharge.

The study will assess changes in self-efficacy, quality of recovery, and selected clinical outcomes to compare recovery between participants who receive the recovery-promoting program and those who receive standard care.

DETAILED DESCRIPTION:
Coronary artery bypass graft (CABG) surgery is a standard treatment for patients with advanced coronary artery disease. Although surgical outcomes have improved, patients frequently experience challenges during postoperative recovery, including reduced physical capacity, delayed functional recovery, psychological distress, and difficulties in self-management after hospital discharge. These challenges may contribute to prolonged recovery and suboptimal clinical outcomes.

Evidence-based approaches such as Cardiac Rehabilitation (CR) and Enhanced Recovery After Cardiac Surgery (ERAS) have been shown to support postoperative recovery. However, in routine clinical practice, the application of these approaches is often fragmented, and continuity of care after discharge remains limited. In particular, patients may receive insufficient guidance and support to enhance self-efficacy and confidence in managing recovery at home.

This study aims to evaluate the effects of a recovery-promoting program on self-efficacy, quality of recovery, and clinical outcomes in patients undergoing CABG surgery. The recovery-promoting program integrates key components of CR and ERAS principles and is delivered by nurses using a structured approach. The intervention includes pre-discharge education, guidance on postoperative activity and symptom management, and follow-up support after discharge through a tele-nursing platform. This approach is designed to enhance patients' engagement in recovery and support continuity of care beyond hospital discharge.

A quasi-experimental design is used to compare outcomes between patients receiving standard postoperative care and those receiving the recovery-promoting program in addition to standard care. Eligible patients are assigned to either a control group or an experimental group according to the study protocol. Data are collected at predefined time points to evaluate changes in self-efficacy, quality of recovery, and selected clinical outcomes.

Self-efficacy and quality of recovery are assessed using validated instruments, while clinical outcomes are obtained from clinical records and routine assessments. The primary focus of the study is to examine differences between groups over time and to explore the potential role of a structured, nurse-led recovery-promoting program in supporting postoperative recovery following CABG surgery.

The findings of this study are expected to contribute to evidence supporting integrated recovery strategies and tele-nursing approaches in postoperative cardiac care and may inform the development of structured nursing interventions to improve recovery outcomes in patients undergoing CABG surgery.

ELIGIBILITY:
Inclusion Criteria:

* Thai patients undergoing elective first-time on-pump coronary artery bypass graft (CABG) surgery alone or combined with valve surgery
* If age >60 years, participants must pass cognitive screening using the 6-Item Cognitive Impairment Test (6-CIT)
* New York Heart Association (NYHA) functional class I-III
* Left ventricular ejection fraction (LVEF) >30%
* Independent in activities of daily living and able to perform the 6-minute walk test (6MWT)

Exclusion Criteria:

* Severe or acute comorbidities within 24 hours prior to surgery (e.g., chronic obstructive pulmonary disease, renal failure, acute myocardial infarction, severe arrhythmia)
* Severe postoperative complications or unstable vital signs (e.g., major bleeding, significant arrhythmia, embolism, need for dialysis, extracorporeal membrane oxygenation)
* Disability or limited ambulation or mobility assessed prior to hospital discharge
* Failure of extubation within 3 days after surgery or requirement for reoperation

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2025-08-22 (Actual); Primary Completion 2026-07-31 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Quality of Recovery after CABG. | up to 8 weeks after surgery
  Quality of recovery will be assessed using the Quality of Recovery-15 (QoR-15) questionnaire, a validated postoperative recovery instrument consisting of 15 items with a total score ranging from 0 to 150. The questionnaire assesses physical comfort, emotional state, psychological support, and physical independence. Higher scores indicate better postoperative recovery.

SECONDARY OUTCOMES:
Self Efficacy | Preoperative, baseline; within 2 weeks prior to surgery and immediately prior to surgery
  Self-efficacy refers to the patient's confidence in managing recovery-related behaviors following coronary artery bypass graft surgery. It will be assessed using the Cardiac Self-Efficacy Scale, a validated questionnaire that measures confidence in managing cardiac symptoms and maintaining functional activities. Total scores range from 0 to 56, with higher scores indicating greater perceived cardiac self-efficacy.
Functional capacity | up to 8 weeks after surgery.
  Functional capacity will be assessed using the 6-Minute Walk Test (6MWT), which measures the distance walked in meters on a flat surface over six minutes. Greater walking distance indicates better functional capacity and postoperative recovery following coronary artery bypass graft surgery.
Pulmonary Function | Baseline (preoperative, at initial patient assessment); perioperative period (at hospital admission); at hospital discharge (postoperative day 7).
  Pulmonary function will be assessed using Peak Expiratory Flow Rate (PEFR), measured in liters per minute. PEFR reflects airway function and respiratory muscle performance and is commonly used to evaluate postoperative pulmonary recovery following coronary artery bypass graft surgery. Higher PEFR values indicate better pulmonary function.
Duration of mechanical ventilation | Perioperative period.
  Duration of mechanical ventilation will be measured as the total number of hours from initiation of postoperative mechanical ventilation until successful extubation. This outcome reflects early postoperative respiratory recovery following coronary artery bypass graft surgery. Shorter duration indicates better respiratory recovery.

CONTACTS AND LOCATIONS:
Locations (1):
- Rajavithi Hospital, Ministry of Public Health, Thailand, Bangkok, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared due to ethical and confidentiality considerations.

REFERENCES:
- [Background] Bandura A. Self-efficacy: toward a unifying theory of behavioral change. Psychol Rev. 1977 Mar;84(2):191-215. doi: 10.1037//0033-295x.84.2.191. No abstract available. PMID 847061
- [Background] Narayanan LT, Hamid SRGS. Incentive spirometry inspiratory capacity changes and predictors after open heart surgery: a 5-day prospective study. Med J Malaysia. 2020 May;75(3):226-234. PMID 32467537
- [Background] Brown TM, Pack QR, Aberegg E, Brewer LC, Ford YR, Forman DE, Gathright EC, Khadanga S, Ozemek C, Thomas RJ; American Heart Association Exercise, Cardiac Rehabilitation and Secondary Prevention Committee of the Council on Clinical Cardiology; Council on Cardiovascular and Stroke Nursing; Council on Lifestyle and Cardiometabolic Health; and Council on Quality of Care and Outcomes Research. Core Components of Cardiac Rehabilitation Programs: 2024 Update: A Scientific Statement From the American Heart Association and the American Association of Cardiovascular and Pulmonary Rehabilitation. Circulation. 2024 Oct 29;150(18):e328-e347. doi: 10.1161/CIR.0000000000001289. Epub 2024 Sep 24. PMID 39315436
- [Background] Yang L, Kaye AD, Venakatesh AG, Green MS, Asgarian CD, Luedi MM, Liu H. Enhanced Recovery after Cardiac Surgery: An Update on Clinical Implications. Int Anesthesiol Clin. 2017 Fall;55(4):148-162. doi: 10.1097/AIA.0000000000000168. No abstract available. PMID 28901988
- [Background] McConnell G, Woltz P, Bradford WT, Ledford JE, Williams JB. Enhanced recovery after cardiac surgery program to improve patient outcomes. Nursing. 2018 Nov;48(11):24-31. doi: 10.1097/01.NURSE.0000546453.18005.3f. PMID 30286030
- [Background] Akowuah EF, Wagnild JM, Bardgett M, Prichard JG, Mathias A, Harrison SL, Ogundimu EO, Hancock HC, Maier RH; PREPs Trial investigators. A randomised controlled trial of prehabilitation in patients undergoing elective cardiac surgery. Anaesthesia. 2023 Sep;78(9):1120-1128. doi: 10.1111/anae.16072. Epub 2023 Jul 4. PMID 37402352
- [Background] Gibbison B, Pufulete M. Prehabilitation before cardiac surgery. Br J Anaesth. 2025 Jan;134(1):5-7. doi: 10.1016/j.bja.2024.11.001. Epub 2024 Nov 26. PMID 39603851
- [Background] Steinmetz C, Bjarnason-Wehrens B, Walther T, Schaffland TF, Walther C. Efficacy of Prehabilitation Before Cardiac Surgery: A Systematic Review and Meta-analysis. Am J Phys Med Rehabil. 2023 Apr 1;102(4):323-330. doi: 10.1097/PHM.0000000000002097. Epub 2022 Sep 23. PMID 36149383
- [Background] Kanejima Y, Shimogai T, Kitamura M, Ishihara K, Izawa KP. Effect of Early Mobilization on Physical Function in Patients after Cardiac Surgery: A Systematic Review and Meta-Analysis. Int J Environ Res Public Health. 2020 Sep 28;17(19):7091. doi: 10.3390/ijerph17197091. PMID 32998202
- [Background] Chen B, Xie G, Lin Y, Chen L, Lin Z, You X, Xie X, Dong D, Zheng X, Li D, Lin W. A systematic review and meta-analysis of the effects of early mobilization therapy in patients after cardiac surgery. Medicine (Baltimore). 2021 Apr 16;100(15):e25314. doi: 10.1097/MD.0000000000025314. PMID 33847630
- [Background] Lapin IP. ["Blank controls" (the complete simulation of the experiment): a comparison of different groups of "control" mice by their indices of spontaneous motor activity]. Zh Vyssh Nerv Deiat Im I P Pavlova. 1996 Sep-Oct;46(5):957-60. No abstract available. Russian. PMID 9054150
- [Background] Zhang Y, Chong JH, Harky A. Enhanced recovery after cardiac surgery and its impact on outcomes: A systematic review. Perfusion. 2022 Mar;37(2):162-174. doi: 10.1177/0267659121988957. Epub 2021 Jan 19. PMID 33468017